CLINICAL TRIAL: NCT00064259
Title: A Phase I/II Study of Oblimersen in Combination With Cisplatin and Fluorouracil in Patients With Advanced Esophageal, Gastro-Esophageal Junction and Gastric Cancer
Brief Title: A Phase I/II Study of Oblimersen Plus Cisplatin and Fluorouracil in Gastric & Esophageal Junction Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Discontinued development of G3139 (oblimersen)
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03134; 02-66 (Other: Montefiore Medical Center); N01CM62204 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-01

CONDITIONS: Adenocarcinoma of the Esophagus; Adenocarcinoma of the Gastroesophageal Junction; Diffuse Adenocarcinoma of the Stomach; Intestinal Adenocarcinoma of the Stomach; Mixed Adenocarcinoma of the Stomach; Recurrent Esophageal Cancer; Recurrent Gastric Cancer; Squamous Cell Carcinoma of the Esophagus; Stage III Esophageal Cancer; Stage IIIA Gastric Cancer; Stage IIIB Gastric Cancer; Stage IIIC Gastric Cancer; Stage IV Esophageal Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms; Stomach Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — oblimersen; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (oblimersen sodium) (Experimental): Phase I: Patients receive oblimersen IV continuously on days 1-7, fluorouracil IV continuously on days 4-8, and cisplatin IV on day 4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 12 patients are treated at the MTD.
  Phase II: Patients receive treatment as in phase I with oblimersen at the MTD.
  Interventions: Biological: oblimersen sodium; Drug: cisplatin; Drug: fluorouracil

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU

SUMMARY:
Drugs used in chemotherapy such as cisplatin and fluorouracil use different ways to stop tumor cells from dividing so they stop growing or die. Oblimersen may increase the effectiveness of chemotherapy by making tumor cells more sensitive to the drugs. This phase I/II trial is studying the side effects and best dose of oblimersen when given with cisplatin and fluorouracil and to see how well they work in treating patients with locally advanced, recurrent, or metastatic cancer of the esophagus, gastroesophageal junction, or stomach.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The escalation portion of the study will determine the MTD of G3139/Cisplatin and will help determine the toxicities of this combination.

II. Once the MTD is determined, an additional 12 patients will be enrolled in order to obtain a set of tumor biopsies for microarray analysis.

SECONDARY OBJECTIVES:

I. The collection of additional toxicity data for this combination

OUTLINE: This is a pilot, multicenter, dose-escalation study of oblimersen.

Phase I: Patients receive oblimersen IV continuously on days 1-7, fluorouracil IV continuously on days 4-8, and cisplatin IV on day 4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 12 patients are treated at the MTD.

Phase II: Patients receive treatment as in phase I with oblimersen at the MTD.

PROJECTED ACCRUAL: Approximately 37-97 patients (3-36 for phase I and 34-67 for phase II) will be accrued for this study within 15-18 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the esophagus, gastro- esophageal junction, or stomach; patients with squamous cell carcinoma of the esophagus will also be eligible, patients must have locally advanced, recurrent or metastatic disease, not amenable to complete surgical resection or definitive radiation therapy
* Measurable and/or evaluable disease
* May have had prior surgery, radiation therapy, combined modality chemo- radiation, or at most one prior chemotherapy regimen for advanced, recurrent or metastatic disease;
* Life expectancy of greater than 12 weeks
* ECOG performance status =<2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* Creatinine =< 1.5 OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Ability to understand and the willingness to sign a written informed consent document
* Patients with accessible tumors are obliged to participate in biopsies 1 and 2; accessible tumors are defined as tumors reachable by EGD, or metastases, which, in the opinion of the treating physician can be biopsied with commonly utilized biopsy methods (such as CT guided biopsy); biopsy #3 on day 6 is optional; patients who do not have have accessible tumor tissue may participate in the study if at least one tumor deposit is measurable

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 21 days (6 weeks for nitrosoureas or mitomycin C, two weeks if prior treatment was a weekly regimen) prior to entering the study or those who have not recovered from adverse events (grade 2 or worse) due to agents administered earlier
* Patients who have had photodynamic therapy within 4 weeks of proposed study entry will be excluded; patients will be allowed to receive concurrent photodynamic therapy for obstruction untreatable by stent, laser, or dilation; patients who do require concurrent photodynamic therapy and who are participating in the serial biopsy portion of the study must wait until after cycle 1 and its biopsies are completed
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to anti- sense oligonucleotides, cisplatin, fluorouracil or other agents used in the study
* Patients may not have received G3139 previously
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because G3139 is an anti- sense oligonucleotide agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with G3139, breastfeeding should be discontinued if the mother is treated with G3139; these potential risks may also apply to other agents used in this study
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with G3139 or other agents administered during the study; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kaubisch, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Result] Raab R, Sparano JA, Ocean AJ, Christos P, Ramirez M, Vinciguerra V, Kaubisch A. A phase I trial of oblimersen sodium in combination with cisplatin and 5-fluorouracil in patients with advanced esophageal, gastroesophageal junction, and gastric carcinoma. Am J Clin Oncol. 2010 Feb;33(1):61-5. doi: 10.1097/COC.0b013e3181a31ad0. PMID 19738454

RESULTS

PARTICIPANT FLOW:
Groups:
- Oblimersen 3 mg/kg/d +Cisplatin 100 mg/m2 +5-FU 1000 mg/m2: Patients received oblimersen as a continuous intravenous infusion (CIVI) on days 1 to 7 at 3 mg/kg/d in combination with CIVI 5-FU 1000 mg/m2/d on days 4 to 7 and cisplatin 100 mg/m2 on day 4.
- Oblimersen 3 mg/kg/d +Cisplatin 75 mg/m2 +5-FU 750 mg/m2: Patients received oblimersen as a continuous intravenous infusion (CIVI) on days 1 to 7 at 3 mg/kg/d in combination with CIVI 5-FU 750 mg/m2/d on days 4 to 7 and cisplatin 75 mg/m2 on day 4.
- Oblimersen 5 mg/kg/d +Cisplatin 75 mg/m2 +5-FU 750 mg/m2: Patients received oblimersen as a continuous intravenous infusion (CIVI) on days 1 to 7 at 5 mg/kg/d in combination with CIVI 5-FU 750 mg/m2/d on days 4 to 7 and cisplatin 75 mg/m2 on day 4.
- Oblimersen 7 mg/kg/d +Cisplatin 75 mg/m2 +5-FU 750 mg/m2: Patients received oblimersen as a continuous intravenous infusion (CIVI) on days 1 to 7 at 7 mg/kg/d in combination with CIVI 5-FU 750 mg/m2/d on days 4 to 7 and cisplatin 75 mg/m2 on day 4.
Period: Overall Study
Arm/Group | Oblimersen 3 mg/kg/d +Cisplatin 100 mg/m2 +5-FU 1000 mg/m2 | Oblimersen 3 mg/kg/d +Cisplatin 75 mg/m2 +5-FU 750 mg/m2 | Oblimersen 5 mg/kg/d +Cisplatin 75 mg/m2 +5-FU 750 mg/m2 | Oblimersen 7 mg/kg/d +Cisplatin 75 mg/m2 +5-FU 750 mg/m2
Started | 4 | 4 | 6 | 1
Completed | 3 | 4 | 6 | 0
Not Completed | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Total number of participants at different dose levels of Oblimersen (3, 5, or 7 mg/kg/d) in combination with 5-FU (1000 mg/m2/d or 750 mg/m2/d) and Cisplatin (100 mg/m2 or 75 mg/m2)
Groups:
- Oblimersen + Cisplatin + 5-FU: Oblimersen dose levels (3, 5, or 7 mg/kg/d) on days 1 to 7 in combination with 5-FU (1000 mg/m2/d or 750 mg/m2/d) on days 4 to 7 and Cisplatin (100 mg/m2 or 75 mg/m2) on day 4.
Arm/Group | Oblimersen + Cisplatin + 5-FU
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 55.0 [36 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Oblimersen in Combination With Cisplatin and 5-FU
Description: Adverse events were evaluated according to the National Cancer Institute Common Toxicity Criteria (version 2.0). DLT was defined as grade 3 to 4 hematologic toxicity lasting more than 1 week after 5-FU/cisplatin, grade 3 to 4 nausea or vomiting occurring later than 11 days after cisplatin, grade 3 to 4 diarrhea occurring later than 10 days after 5-FU, and grade 3 to 4 mucositis at the beginning of the next cycle.
Time Frame: 21 days
Measure: Number; unit: mg/kg/d
Arm/Group | Oblimersen + Cisplatin + 5-FU
Number analyzed (Participants) | 15
mg/kg/d | 5

2. Secondary Outcome: Microarray Data
Description: This will be primarily descriptive, and will seek to compare patterns of gene expression pre- and post-treatment.
Time Frame: Up to 12 weeks
Population: Outcome was not analysed. No patients had samples obtained for microarray analysis.
Groups:
- Treatment (Oblimersen Sodium): Phase I: Patients receive oblimersen IV continuously on days 1-7, fluorouracil IV continuously on days 4-8, and cisplatin IV on day 4. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of oblimersen until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 12 patients are treated at the MTD.
  Phase II: Patients receive treatment as in phase I with oblimersen at the MTD.
  oblimersen sodium: Given IV
  cisplatin: Given IV
  fluorouracil: Given IV
Arm/Group | Treatment (Oblimersen Sodium)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Oblimersen + Cisplatin + 5-FU
Serious Adverse Events (participants affected / at risk) | 8/15
Other Adverse Events (participants affected / at risk) | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oblimersen + Cisplatin + 5-FU (N=15)
Neutropenia (Blood and lymphatic system disorders) | 5
Anemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Infection (Infections and infestations) | 3
Vomiting (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Transaminase elevation (Hepatobiliary disorders) | 1
Alkaline phosphatase (Hepatobiliary disorders) | 1
Creatinine (Renal and urinary disorders) | 1
Ureteral obstruction (Renal and urinary disorders) | 1
Fatigue (General disorders) | 2
Dizziness (General disorders) | 2
Vascular/Thrombosis (Vascular disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Sensory neuropathy (Nervous system disorders) | 1
Motor neuropathy (Nervous system disorders) | 1
Pleural effusion (General disorders) | 1
Ascites (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oblimersen + Cisplatin + 5-FU (N=15)
Neutropenia (Blood and lymphatic system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Mucositis (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Alkaline phosphatase (Hepatobiliary disorders) | 2
Weight loss (General disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 3
Dizziness (General disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Peripheral edema (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less